CLINICAL TRIAL: NCT00747799
Title: Phase II Study of Combination of Sorafenib With Cisplatin and 5-fluorouracil as First-line Treatment of Recurrence After Radiotherapy Patients Who Are Failure of Radiotherapy in Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC)
Brief Title: Study of Combination of Sorafenib With Cisplatin and 5-fluorouracil as First-line Treatment of Recurrence After Radiotherapy Patients Who Failed With Radiotherapy in Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Profressor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAY43-9006-2008003
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2011-11

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: recurrent or metastatic Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Recurrence | interventions — Sorafenib; Cisplatin; Fluorouracil

ARMS (1):
- 1 (Experimental): Sorafenib with Cisplatin and 5-fluorouracil as first-line treatment of recurrence after radiotherapy patients who failed with radiotherapy in recurrent or metastatic nasopharyngeal carcinoma (NPC)
  Interventions: Drug: Sorafenib plus Cisplatin and 5-fluorouracil

INTERVENTIONS:
Drug: Sorafenib plus Cisplatin and 5-fluorouracil — Sorafenib with Cisplatin and 5-fluorouracil as first-line treatment of recurrence after radiotherapy patients who failed with radiotherapy in recurrent or metastatic nasopharyngeal carcinoma (NPC)
  * Sorafenib 400 mg bid per daily . Every 21-day cycles.
  * Cisplatin 80 mg/m2 day d1, every 21 days cycle.
  * 5-fluorouracil 1000 mg/m2 day CIV 4days, repeat 21-day cycles

SUMMARY:
This study is a phase II clinical study. Recurrence after radiotherapy patients who are failure of radiotherapy in recurrent or metastatic nasopharyngeal carcinoma (NPC) were treated by cisplatin and 5-fluorouracil with Sorafenib as first-line treatment. The objective response(complete response (CR) + partial response (PR)), Disease Control Rate , safety profile, tolerability will be evaluated according to World Health Organization (WHO) criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. ECOG Performance Status of 0 or 1
3. Life expectancy of at least 12 weeks
4. Pathologically confirmed nasopharyngeal carcinoma
5. Experience of treatment failure with radiotherapy for recurrent or metastatic NPC
6. More than 3 weeks must have elapsed since previous radiotherapy
7. Biomarkers measuring including pERK, EGFR of original diagnostic paraffin-embedded tumor samples; VEGF of pre-dose and post-dose plasma samples.
8. Subjects with at least one (for RECIST) measurable lesion (Tumor lesions that are situated in a previously irradiated area could not be considered measurable)
9. Adequate bone marrow, liver and renal functions as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

   * Hemoglobin > 9.0 g/dl
   * Absolute neutrophil count (ANC) > 1,500/mm3
   * Platelet count > 100,000/μl
   * Total bilirubin < 1.5 times the upper limit of normal
   * ALT and AST < 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer), Alkaline phosphatase < 4 x ULN ,PT-INR/PTT < 1.5 x upper limit of normal, Serum creatinine < 1.5 x upper limit of normal
10. Signed and dated informed consent before the start of specific protocol procedures

Exclusion Criteria:

1. History of cardiac disease: congestive heart failure > NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension.
2. History of HIV infection
3. Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
4. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
5. History of organ allograft the organ allograft may be allowed as protocol specific.
6. Patients with evidence or history of bleeding diatheses
7. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
8. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial.
9. Patients unable to swallow oral medications
10. Prior use of farnesyl transferase, Raf kinase, or MEK inhibitors
11. Investigational drug therapy outside of this trial during or within 4 weeks of study entry
12. Prior exposure to the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate (CR+PR) | January 2009 to May 2011
  In the ITT analysis(n=54), the ORR reached 77.8%: one patient (1.9%) experienced CR; 41 (75.9%), PR.

SECONDARY OUTCOMES:
Disease control rate | January 2009 to May 2011
  The disease control rate (DCR) was 90.8%.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center of Sun-Yat Sen University, Guangzhou, Guangdong, China